CLINICAL TRIAL: NCT04758546
Title: Customizing Spontaneous Breathing Trial After Aggressive Readiness Criteria Hastens Weaning in Low and Intermediate Risk Patients With Prevention: A Randomized Trial (SPEED-UP Trial).
Brief Title: Speeding the Weaning up: Aggressive Screening Criteria and Higher Minimal Ventilatory Settings.
Acronym: SPEED-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gonzalo Hernandez Martinez (Other)
Responsible Party: Sponsor-Investigator, Gonzalo Hernandez Martinez, MD, PhD, Hospital Virgen de la Salud
Organization: Hospital Virgen de la Salud (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 7/10/2020 Nº 10
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Weaning Failure
MeSH Terms: interventions — Weaning

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aggressive screening criteria + high minimal ventilatory settings (Experimental)
  Interventions: Diagnostic Test: Screening criteria for weaning and minimal ventilatory settings for spontaneous breathing trial
- Aggressive screening criteria + low minimal ventilatory settings (Experimental)
  Interventions: Diagnostic Test: Screening criteria for weaning and minimal ventilatory settings for spontaneous breathing trial
- Conservative screening criteria + high minimal ventilatory settings (Experimental)
  Interventions: Diagnostic Test: Screening criteria for weaning and minimal ventilatory settings for spontaneous breathing trial
- Conservative screening criteria + low minimal ventilatory settings (Active Comparator)
  Interventions: Diagnostic Test: Screening criteria for weaning and minimal ventilatory settings for spontaneous breathing trial

INTERVENTIONS:
Diagnostic Test: Screening criteria for weaning and minimal ventilatory settings for spontaneous breathing trial — Aggressive screening criteria: Walsh Conservative screening criteria: Boles High minimal ventilatory settings: pressure Support 8 + positive end-expiratory pressure 5 Low minimal ventilatory settings: pressure support 5

SUMMARY:
Hypothesis:

1. In patients with less than 4 high risk factors for reintubation excluding body mass index >30 and hypercapnia during the spontaneous breathing trial (SBT) (low and intermediate risk for extubation failure), who receive preventive therapy with high flow nasal cannula (HFNC), the use of SBT with "HIGH minimal ventilator settings" (PS 8 + PEEP 5 cm H2O Vs PS 5 + PEEP 0 cm H2O), increase the proportion of patients with simple weaning (extubation after the first SBT).
2. In patients with low and intermediate risk for extubation failure, who receive preventive therapy with HFNC, the use of Walsh screening criteria reduces the mechanical ventilation time compared with the use of Boles criteria.

Study design: This is a multicenter randomized open trial with 4 arms.

1. Screening with PaO2/FiO2 > 180 and PEEP ≤ 10cm H2O; SBT with "HIGH minimal ventilator settings" (PS 8 + PEEP 5 cm H2O).
2. Screening with PaO2/FiO2 > 180 and PEEP ≤ 10 cm H2O; SBT with "LOW minimal ventilator settings" (PS 5 + PEEP 0 cm H2O).
3. Screening with PaO2/FiO2 ≥ 150 and PEEP ≤ 8 cm H2O; SBT with "HIGH minimal ventilator settings" (PS 8 + PEEP 5 cm H2O).
4. Screening with PaO2/FiO2 ≥ 150 and PEEP ≤ 8 cm H2O; SBT with "LOW minimal ventilator settings" (PS 5 + PEEP 0 cm H2O).

Primary Outcome Measure:

1. - Percentage of first spontaneous breathing trial tolerated.
2. - Time on mechanical ventilation.

DETAILED DESCRIPTION:
Discontinuation of mechanical ventilation is a three-step process including:

1. - Readiness testing.

   It evaluates the criteria to determine whether a patient might be able to be successfully and safety weaned from mechanical ventilation. The detection of readiness to try a spontaneous breathing test has controversial questions, in special concerning to oxygenation. From a conservative to an aggressive criteria we can list:
   1. PaO2/FiO2 > 200 on PEEP ≤ 5 cm H2O (Esteban et al, 1999).
   2. PaO2/FiO2 ≥ 150 on PEEP ≤ 8 cm H2O (Boles et al, 2007).
   3. PaO2/FiO2 > 180 on PEEP ≤ 10 cm H2O (Walsh et al, 2004). We will compare Walsh and Boles in their different considerations for oxygenation criteria. Since Walsh criteria require a higher level of PEEP we understand that this criteria is more aggressive and in this way it allow to an early detection of readiness to SBT, but there is not any evidence of this statement.
2. - Spontaneous breathing trial (SBT). It tries to simulate (but not only) post-extubation work of breathing to promptly determine the time to extubation. There is also disparity about SBT minimal ventilator settings:

   1. Inspiratory pressure with a range between automatic tube compensation (ATC) and inspiratory pressure of 5 - 8 cm H2O. Theoretically, if we use a higher support pressure during SBT it would be easier to pass the test. One could think that this may rise the risk of reintubation but there are various trials that have not confirmed this assumption.
   2. Guidelines does not make any recommendation about expiratory pressurization, although the trials conducted use levels of Positive End-Expiratory Pressure (PEEP), between 0 and 5 cm H2O.
   3. Furthermore, we consider that "minimal ventilator settings" must be adjusted to additional parameters not previously considered, like preventive therapy applied after the extubation.
   4. All spontaneous breathing trials will last 30 minutes.
3. - Extubation follow-up care. Therapies targeted to prevent post-extubation respiratory failure like high flow nasal cannula (HFNC), noninvasive ventilation (NIV) and respiratory physiotherapy for improving airway clearance, have been proposed.

The variability of preventive therapies and its settings generate different "minimal ventilator settings".

In view of all that has been set out above, there are two essential points that has not been analyzed as far we understand:

1. The different screening criteria available have not been compared with each other about allowing early detection of readiness, even less with the individual risk of postextubation failure and still less with the preventive therapy that would be applied for each group.
2. The different inspiratory support pressure as well as PEEP level, have not been compared with other different values, even less with the individual risk of postextubation failure and still less with the preventive therapy that would be applied for each group.

The detailed weaning criteria include the following:

* Clinical evaluation:

  * Adequate cough reflex and good clearance of respiratory secretions.
  * Resolution or stabilization of the initial reason for intubation.
  * Patient awake with RASS between +1 and -2 according the Richmond Assessment Sedation Scale (RASS).
* Data evaluation:

  * Cardiovascular stability with minimal or no need of vasopressors (HR ≤ 140 lpm, blood systolic pressure between 90-160 mmHg with minimal or no need of vasopressors and without increase in the last 24 hours).
  * Successful oxygenation defined by SpO2 >90% on FiO2 ≤ 40% or PaO2/FiO2

    ≥150 with PEEP up to ≤8 cmH2O (Boles et al, 2007) or PaO2/FiO2 >180 con PEEP ≤10 cm H2O (Walsh et al, 2004).
  * Respiratory rate ≤35 bpm without respiratory acidosis.
  * Hemoglobin >7g/dL.
  * Temperature between 36-38,5ºC.
  * Blood potassium between 3-5 mmol/L.
  * Blood sodium between 128-150 mmol/L.

Detailed definition of high risk factors for extubation failure: age older than 65 years; heart failure as the primary indication for mechanical ventilation; moderate to severe chronic obstructive pulmonary disease; an Acute Physiology and Chronic Health Evaluation II (APACHE II) score higher than 12 on extubation day; body mass index of more than 30 (calculated as weight in kilograms divided by height in meters squared); airway patency problems, including high risk of developing laryngeal edema; inability to deal with respiratory secretions (inadequate cough reflex or suctioning >2 times within 8 hours before extubation); difficult or prolonged weaning, in brief, a patient failing the first attempt at disconnection from mechanical ventilation; 2 or more comorbidities defined with Charlson score; and mechanical ventilation for more than 7 days.

The detailed risk categories are the following:

* Low risk: Patients without risk factors who benefit from HFNC.
* Intermediate risk: Patients with 1 to 3 risk factors excluding obese (BMI >30 Kg/m2) and those who develop hypercapnia during the SBT, that can benefit from HFNC.
* High risk: Obese (BMI >30 Kg/m2) and patients with 4 or more risk factors including hypercapnia during the SBT. This group may benefit from prevention with NIV.

Sample size estimation:

* Basal parameters in low risk patients treated with post-extubation HFNC: estimated 30% of the entire population. Reintubation rate 4.9% and 1(1-3) days on mechanical ventilation. Estimated reduction in the intervention group: 1 day in the 25% of the patients.
* Basal parameters in intermediate risk patients treated with HFNC: estimated 70% of the entire population. Reintubation rate 12.24% and 4 (2 - 9) days on mechanical ventilation. Estimated reduction 1 day in the 33% of the patients).

Calculated standard deviation 3.5 days. CI 95% and power 80%, loss rate 10%, and one-tail analysis: 260 patients per group.

Simple randomization immediately after finishing the spontaneous breathing trial. An intention to treat analysis will be performed.

Detailed HFNC treatment: High-flow oxygen (Optiflow, Fisher and Paykel Healthcare) will be applied immediately after extubation through specific nasal cannula. Flow will be initially set at 10 L/min and titrated upwards in 5-L/min steps until patients experience discomfort. Temperature will be initially set to 37°C, unless reported too hot by patients, and FIO2 will be regularly adjusted to the target peripheral capillary oxygen saturation (SPO2) of greater than 92%. After 48 hours, high-flow will be stopped and, if necessary, patients will receive conventional oxygen therapy.

Criteria for spontaneous breathing trial failure are: agitation, anxiety, depressed mental status, diaphoresis, cyanosis, evidence of increasing respiratory effort, increased accessory muscle activity, facial signs of distress, dyspnea, PaO2 lower than 60 mmHg or SpO2 lower than 90% on inspired fraction of oxygen higher than .5, PaCO2 higher than 50 mmHg or increased more than 8 mmHg from baseline value, arterial pH lower than 7.32 or decreased more than .07 from baseline value, respiratory rate higher than 35 breaths per minute or increased more than 50% from baseline value, heart rate higher than 140 beats per minute or increased more than 20% from baseline value, systolic arterial pressure higher than 180 mmHg or increased more than 20% from baseline value, systolic arterial pressure lower than 90 mmHg, or cardiac arrhythmias.

Patients who tolerate the spontaneous breathing trial will be reconnected with the previous ventilator settings for rest and clinical evaluation of airway patency, respiratory secretions, and upper airway obstruction before extubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation for more than 24 hours with >= positive end-expiratory pressure 10.
* Patients with up to three high risk factors for extubation failure excluding hypercapnia during the spontaneous breathing trial and obese patients (BMI >30).
* Patients fulfilling weaning criteria expected to have a spontaneous breathing trial in the following 24 hours.
* Patients expected to be prevented with high-flow oxygen therapy after extubation.

Exclusion Criteria:

* <18 years old.
* Pregnant women.
* Tracheostomized patients.
* Accidental or self-extubated patients.
* Obese (BMI >30) or hypercapnic patients during the spontaneous breathing trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of first spontaneous breathing trial tolerated | 1 month after intubation
Time on mechanical ventilation | 1 month after intubation

SECONDARY OUTCOMES:
Reintubation rate | 7 days after extubation
Post-extubation respiratory failure rate | 7 days after extubation
ICU and Hospital length of stay | 3 months after ICU and Hospital admission
ICU and Hospital mortality rate | 3 months after ICU and Hospital admission
Sepsis and multiorgan failure rate | 3 months after ICU and Hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Hernandez, Study Chair — University Hospital Virgen de la Salud
Locations (1):
- Hospital Virgen de la Salud, Toledo, Castille-La Mancha, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hernandez Martinez G, Rodriguez P, Soto J, Caritg O, Castellvi-Font A, Mariblanca B, Garcia AM, Colinas L, Anon JM, Parrilla-Gomez FJ, Silva-Obregon JA, Masclans JR, Propin A, Cuadra A, Dalorzo MG, Rialp G, Suarez-Sipmann F, Roca O. Effect of aggressive vs conservative screening and confirmatory test on time to extubation among patients at low or intermediate risk: a randomized clinical trial. Intensive Care Med. 2024 Feb;50(2):258-267. doi: 10.1007/s00134-024-07330-w. Epub 2024 Feb 14. PMID 38353714